CLINICAL TRIAL: NCT02925520
Title: Expanded Access Use of Omegaven® in the Treatment of Parenteral Nutrition Induced Liver Injury in Children
Status: No longer available | Type: Expanded Access
Sponsor: Cook Children's Health Care System (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-059
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Parenteral Nutrition-Associated Liver Disease
Keywords: Cholestasis
MeSH Terms: conditions — Cholestasis | interventions — fish oil triglycerides; Fish Oils

INTERVENTIONS:
Drug: Omegaven — Therapy with Omegaven will be provided at a dose of 1 gm/kg/day infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition. Parenteral fat emulsion (Intralipid) will be administered only if necessary to administer adequate calories during Omegaven therapy. The same standards of care provided to all patients receiving parenteral nutrition solution will be followed.
  Home Use of Omegaven:
  The Omegaven dose for home use will be the same as that used while in the hospital: 1 gm/kg/day. As with the inpatient part of the protocol, this is a maximum dose and may be decreased at the discretion of the provider.
  Other Names: Fish oil

SUMMARY:
This is an expanded access study to assess the safety profile and changes in serum direct bilirubin levels in infants with PN associated cholestasis. Eligible patients will receive therapy with Omegaven on an expanded access basis by method of continuous infusion. Omegaven will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition. The same standards of care provided to all patients receiving parenteral nutrition solution will be followed.

DETAILED DESCRIPTION:
This expanded access protocol provides a mechanism for critically ill infants with parenteral nutrition-associated liver disease (PNALD) to receive Omegaven for compassionate use situations for which there are no satisfactory alternative treatments.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 4 weeks (28 days) old and less then 5 years of age
* Diagnosis of PNALD as defined by serum direct bilirubin greater than 2 mg/dL on 2 consecutive occasions
* Expected to require intravenous nutrition for at least an additional 28 days
* Have been PN-dependent for at least four weeks prior to planned Omegaven initiation
* PN-dependent and unable to meet nutritional requirements by enteral means
* Have failed standard therapies to prevent progression of PNALD
* Hospitalized at time of Omegaven initiation

Exclusion Criteria:

* Have a congenitally lethal condition (e.g. Trisomy 13).
* Have evidence of a viral hepatitis or primary liver disease as the primary etiology of their cholestasis.
* Have other health problems such that survival is extremely unlikely even if the infant's cholestasis improves.
* Have been in another clinical trial within 30 days prior to enrollment or received an investigational drug within 30 days prior to enrollment or scheduled to receive an investigational drug other than Omegaven during the study period.
* Severe and/or unstable concomitant systemic disease such as complex congenital cardiac disease, renal failure, autoimmune disease, sepsis, inborn error of metabolism, genetic liver disease
* Bleeding disorder
* Biochemical disturbance with potential of worsening with proposed treatment, e.g. persistent hyperglycemia, hypertriglyceridemia, hypercalcemia.

Ages: 4 Weeks to 5 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Bankole O Osuntokun, MD, MS, Principal Investigator — Cook Children's Medical Center
Locations (1):
- Cook Children's Medical Center, Fort Worth, Texas, United States

REFERENCES:
- [Background] Dudrick SJ, Wilmore DW, Vars HM, Rhoads JE. Long-term total parenteral nutrition with growth, development, and positive nitrogen balance. 1968. Nutr Hosp. 2001 Nov-Dec;16(6):287-92; discussion 286-7. No abstract available. PMID 11845800
- [Background] Wilmore DW, Dudrick SJ. Growth and development of an infant receiving all nutrients exclusively by vein. JAMA. 1968 Mar 4;203(10):860-4. No abstract available. PMID 4965871
- [Background] Mullick FG, Moran CA, Ishak KG. Total parenteral nutrition: a histopathologic analysis of the liver changes in 20 children. Mod Pathol. 1994 Feb;7(2):190-4. PMID 8008742
- [Background] Freund HR. Abnormalities of liver function and hepatic damage associated with total parenteral nutrition. Nutrition. 1991 Jan-Feb;7(1):1-5; discussion 5-6. PMID 1802177
- [Background] Beath SV, Davies P, Papadopoulou A, Khan AR, Buick RG, Corkery JJ, Gornall P, Booth IW. Parenteral nutrition-related cholestasis in postsurgical neonates: multivariate analysis of risk factors. J Pediatr Surg. 1996 Apr;31(4):604-6. doi: 10.1016/s0022-3468(96)90507-2. PMID 8801324
- [Background] Greenberg GR, Wolman SL, Christofides ND, Bloom SR, Jeejeebhoy KN. Effect of total parenteral nutrition on gut hormone release in humans. Gastroenterology. 1981 May;80(5 pt 1):988-93. No abstract available. PMID 6781979
- [Background] Yeh SL, Chen WJ, Huang PC. Effects of L-glutamine on induced hepatosteatosis in rats receiving total parenteral nutrition. J Formos Med Assoc. 1995 Oct;94(10):593-9. PMID 8527958
- [Background] Kubota A, Yonekura T, Hoki M, Oyanagi H, Kawahara H, Yagi M, Imura K, Iiboshi Y, Wasa K, Kamata S, Okada A. Total parenteral nutrition-associated intrahepatic cholestasis in infants: 25 years' experience. J Pediatr Surg. 2000 Jul;35(7):1049-51. doi: 10.1053/jpsu.2000.7769. PMID 10917294
- [Background] Moss RL, Das JB, Ansari G, Raffensperger JG. Hepatobiliary dysfunction during total parenteral nutrition is caused by infusate, not the route of administration. J Pediatr Surg. 1993 Mar;28(3):391-6; discussion 396-7. doi: 10.1016/0022-3468(93)90238-g. PMID 8468653
- [Background] Helms RA, Christensen ML, Mauer EC, Storm MC. Comparison of a pediatric versus standard amino acid formulation in preterm neonates requiring parenteral nutrition. J Pediatr. 1987 Mar;110(3):466-70. doi: 10.1016/s0022-3476(87)80519-x. No abstract available. PMID 3102712
- [Background] Moss RL, Haynes AL, Pastuszyn A, Glew RH. Methionine infusion reproduces liver injury of parenteral nutrition cholestasis. Pediatr Res. 1999 May;45(5 Pt 1):664-8. doi: 10.1203/00006450-199905010-00009. PMID 10231861
- [Background] Meehan JJ, Georgeson KE. Prevention of liver failure in parenteral nutrition-dependent children with short bowel syndrome. J Pediatr Surg. 1997 Mar;32(3):473-5. doi: 10.1016/s0022-3468(97)90609-6. PMID 9094021
- [Background] Whalen GF, Shamberger RC, Perez-Atayde A, Folkman J. A proposed cause for the hepatic dysfunction associated with parenteral nutrition. J Pediatr Surg. 1990 Jun;25(6):622-6. doi: 10.1016/0022-3468(90)90348-d. PMID 2113578
- [Background] Zamir O, Nussbaum MS, Bhadra S, Subbiah MT, Rafferty JF, Fischer JE. Effect of enteral feeding on hepatic steatosis induced by total parenteral nutrition. JPEN J Parenter Enteral Nutr. 1994 Jan-Feb;18(1):20-5. doi: 10.1177/014860719401800120. PMID 8164298
- [Background] Kaminski DL, Adams A, Jellinek M. The effect of hyperalimentation on hepatic lipid content and lipogenic enzyme activity in rats and man. Surgery. 1980 Jul;88(1):93-100. No abstract available. PMID 6104363
- [Background] Hultin M, Carneheim C, Rosenqvist K, Olivecrona T. Intravenous lipid emulsions: removal mechanisms as compared to chylomicrons. J Lipid Res. 1995 Oct;36(10):2174-84. PMID 8576643
- [Background] Qi K, Al-Haideri M, Seo T, Carpentier YA, Deckelbaum RJ. Effects of particle size on blood clearance and tissue uptake of lipid emulsions with different triglyceride compositions. JPEN J Parenter Enteral Nutr. 2003 Jan-Feb;27(1):58-64. doi: 10.1177/014860710302700158. PMID 12549600
- [Background] Nestel PJ. Effects of N-3 fatty acids on lipid metabolism. Annu Rev Nutr. 1990;10:149-67. doi: 10.1146/annurev.nu.10.070190.001053. No abstract available. PMID 2200461
- [Background] Chen WJ, Yeh SL, Huang PC. Effects of fat emulsions with different fatty acid composition on plasma and hepatic lipids in rats receiving total parenteral nutrition. Clin Nutr. 1996 Feb;15(1):24-8. doi: 10.1016/s0261-5614(96)80257-3. PMID 16843991
- [Background] Yeh SL, Chen WJ, Huang PC. Effects of fish oil and safflower oil emulsions on diet-induced hepatic steatosis in rats receiving total parenteral nutrition. Clin Nutr. 1996 Apr;15(2):80-3. doi: 10.1016/s0261-5614(96)80024-0. PMID 16844003
- [Background] Kinsella JE, Lokesh B, Broughton S, Whelan J. Dietary polyunsaturated fatty acids and eicosanoids: potential effects on the modulation of inflammatory and immune cells: an overview. Nutrition. 1990 Jan-Feb;6(1):24-44; discussion 59-62. No abstract available. PMID 2135755
- [Background] Gura KM, Lee S, Valim C, Zhou J, Kim S, Modi BP, Arsenault DA, Strijbosch RA, Lopes S, Duggan C, Puder M. Safety and efficacy of a fish-oil-based fat emulsion in the treatment of parenteral nutrition-associated liver disease. Pediatrics. 2008 Mar;121(3):e678-86. doi: 10.1542/peds.2007-2248. PMID 18310188
- [Background] Strijbosch RA, Lee S, Arsenault DA, Andersson C, Gura KM, Bistrian BR, Puder M. Fish oil prevents essential fatty acid deficiency and enhances growth: clinical and biochemical implications. Metabolism. 2008 May;57(5):698-707. doi: 10.1016/j.metabol.2008.01.008. PMID 18442636